CLINICAL TRIAL: NCT03999268
Title: Evaluation of Insulin Start Therapy Application With Resources and Training (I-START) to Address Barriers to Insulin Therapy
Brief Title: Insulin Start Therapy Application With Resources and Training
Acronym: I-START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Linda Siminerio, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040017
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Psychological insulin resistance; Diabetes self-management; Mobile application
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention group will receive insulin administration education according to standard procedures plus have access to the I-START app. Over the course of the study period, participants will be able to use I-START as much or as little as they prefer.
  Interventions: Behavioral: I-START; Behavioral: Standard Insulin Administration Education
- Usual Care (Active Comparator): Participants in the usual care group will receive insulin administration education according to standard procedures. They will not have access to the I-START app.
  Interventions: Behavioral: Standard Insulin Administration Education

INTERVENTIONS:
Behavioral: I-START — Designed as a supplementary educational tool for patients on insulin therapy, I-START includes an injection plan to reinforce the knowledge and behaviors that users have been taught by their health care provider. This is done through eight modules created for the benefit of new and experienced insulin users, and those using pens or vial/syringes. The modules address a variety of topics pertinent to insulin therapy, including overcoming psychosocial barriers, injection techniques and best practices, managing hypo- and hyperglycemic events, monitoring blood glucose and troubleshooting and problem solving. At the end of each module, users can self-evaluate their confidence in mastering the information presented. This gives them the ability to move forward into the next module, repeat material already presented and/or save features of the modules that they would like to revisit at another time.
  Arms: Intervention
Behavioral: Standard Insulin Administration Education — Standard best practices for training patients to administer insulin therapy include 1) a thorough patient assessment prior to therapy initiation to address barriers, including evaluation for diminished cognitive capacity or other problem that may impair safe insulin self-administration, and assessment of health literacy and numeracy skills; 2) observation of a patient's injection practice, with re-education provided as needed; 3) use of appropriate language is necessary when teaching injection technique; 4) dose preparation, which includes inspecting the insulin dose for accuracy (following manufacturer instructions); and 5) review of signs, symptoms and treatment of hypoglycemia must be included as a critical component of the training.

SUMMARY:
The purpose of the I-START study is to evaluate an educational phone application (app) designed to support patients with type 2 diabetes (T2DM) by reinforcing the necessary skills needed for insulin administration as part of diabetes self-management.

DETAILED DESCRIPTION:
Despite advances in technology and delivery systems, patients with T2DM continue to be reluctant to begin and adhere to insulin therapy for a variety of reasons. Introducing insulin therapy is particularly problematic during a hospitalization or a brief routine outpatient visit given time and resource constraints. Teaching people to administer an insulin injection requires time and ongoing support. Therefore, this study aims to evaluate an educational phone application designed to support patients with T2DM by reinforcing skills and self-management behaviors needed for insulin administration. Patients with T2DM who are starting insulin or need updated instruction on insulin will be invited to participate in this study to examine the effect of the phone app on psychological barriers to insulin as well as patient and provider satisfaction with and usability of the phone app in both outpatient and hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Able to read and follow study instructions in English (translations will not be provided)
* T2DM requiring the use of prandial and/or long-acting insulin
* Ability to self-administer insulin therapy
* Willing to download the study app on their smartphone
* Able and willing to provide a signed consent
* Able and willing to follow all study procedures

Exclusion Criteria:

* Pregnant (self-reported)
* Participants from the same household participating concurrently
* Use of a smartphone with iOS version 10.0 or lower
* Use of a smartphone with Android OS 5.0 "Lollipop" or lower
* Currently using a continuous subcutaneous insulin infusion device
* Participants with major depression
* Currently or planning to participate in a similar study that would affect the results of this study
* Currently or planning to participate in a clinical study that involves taking a drug, supplement, or use of an investigational drug
* Continued hospitalization or transfer to an assisted living facility
* Any condition the PI or designee deems to pose a risk to the participant in the study (includes anything that may prevent full participation in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in psychological insulin resistance at 2 weeks | 2 weeks
  Psychological insulin resistance will be assessed using the Barriers to Insulin Treatment Questionnaire (BIT), a short instrument that is easy to administer and may be used by both clinicians and researchers (Petrak et al, 2007). The BIT Questionnaire includes 14 items, a total sum score, and the following five subscales: fear of injection and self-testing, expectations regarding positive insulin related outcomes, expected hardship from insulin treatment, stigmatization by insulin injection, and fear of hypoglycemia. Each item is scored on a scale from 1 to 10, which are summed and averaged for total scores; the higher the score, the greater the level of concern.
Change from baseline in psychological insulin resistance at 3 months | 3 months
  Psychological insulin resistance will be assessed using the Barriers to Insulin Treatment Questionnaire (BIT), a short instrument that is easy to administer and may be used by both clinicians and researchers (Petrak et al, 2007). The BIT Questionnaire includes 14 items, a total sum score, and the following five subscales: fear of injection and self-testing, expectations regarding positive insulin related outcomes, expected hardship from insulin treatment, stigmatization by insulin injection, and fear of hypoglycemia. Each item is scored on a scale from 1 to 10, which are summed and averaged for total scores; the higher the score, the greater the level of concern.
Change from baseline in psychological insulin resistance at 6 months | 6 months
  Psychological insulin resistance will be assessed using the Barriers to Insulin Treatment Questionnaire (BIT), a short instrument that is easy to administer and may be used by both clinicians and researchers (Petrak et al, 2007). The BIT Questionnaire includes 14 items, a total sum score, and the following five subscales: fear of injection and self-testing, expectations regarding positive insulin related outcomes, expected hardship from insulin treatment, stigmatization by insulin injection, and fear of hypoglycemia. Each item is scored on a scale from 1 to 10, which are summed and averaged for total scores; the higher the score, the greater the level of concern.

SECONDARY OUTCOMES:
Change from baseline in glycemic control at 3 months | 3 months
  Hemoglobin A1c (HbA1c) will serve as a clinical indicator of glycemic control. HbA1c will serve as the clinical study outcome and measure of glycemic control. HbA1c values will be obtained from the electronic medical record (EMR) system.
Change from baseline in glycemic control at 6 months | 6 months
  Hemoglobin A1c (HbA1c) will serve as a clinical indicator of glycemic control. HbA1c will serve as the clinical study outcome and measure of glycemic control. HbA1c values will be obtained from the electronic medical record (EMR) system.
Change from baseline in medication adherence at 3 months | 3 months
  Medication adherence will be assessed with the 8-item Morisky Medication Adherence Scale (MMAS-8). The scales includes 8 items. Scores can range from 0 to 8; the higher the score, the more adherent the respondent is considered.
Change from baseline in medication adherence at 6 months | 6 months
  Medication adherence will be assessed with the 8-item Morisky Medication Adherence Scale (MMAS-8). Scores can range from 0 to 8; the higher the score, the more adherent the respondent is considered.
Change from baseline in diabetes empowerment at 3 months | 3 months
  Empowerment will be measured using the 8-item Diabetes Empowerment Scale-Short Form (DES-SF), which measures an individual's perceived ability to manage psychosocial aspects of diabetes, assess dissatisfaction and readiness to change self-management plans and set and achieve diabetes goals (Anderson et al, 2000; Anderson et al, 2003). Possible scores are 1 to 5 for each item, summed for a possible total score of 8 to 40. Higher scores indicate greater empowerment.
Change from baseline in diabetes empowerment at 6 months | 6 months
  Empowerment will be measured using the 8-item Diabetes Empowerment Scale-Short Form (DES-SF), which measures an individual's perceived ability to manage psychosocial aspects of diabetes, assess dissatisfaction and readiness to change self-management plans and set and achieve diabetes goals (Anderson et al, 2000; Anderson et al, 2003). Possible scores are 1 to 5 for each item, summed for a possible total score of 8 to 40. Higher scores indicate greater empowerment.
Change from baseline in diabetes distress at 3 months | 3 months
  Diabetes distress will be evaluated with the 17-item Diabetes Distress Scale (DDS17), which assesses four dimensions of distress - emotional, regimen, interpersonal and physician (Polonsky et al, 2005), and has shown a consistent pattern of relationships with HbA1c, diabetes self-efficacy, diet and physical activity in multiple samples of patients with T2DM (Fisher et al, 2012). Individual items are scored from 1 to 6; total scores are the average of all individual item scores; higher scores indicate greater distress.
Change from baseline in diabetes distress at 6 months | 6 months
  Diabetes distress will be evaluated with the 17-item Diabetes Distress Scale (DDS17), which assesses four dimensions of distress - emotional, regimen, interpersonal and physician (Polonsky et al, 2005), and has shown a consistent pattern of relationships with HbA1c, diabetes self-efficacy, diet and physical activity in multiple samples of patients with T2DM (Fisher et al, 2012). Individual items are scored from 1 to 6; total scores are the average of all individual item scores; higher scores indicate greater distress.
Patient Satisfaction | 6 months
  Patient satisfaction will be assessed using the validated Diabetes Medication System Rating Questionnaire-Short Form (DMSRQ-SF) (Peyrot et al, 2014). Items are scored 0 to 100; higher scores equal greater levels of item/construct being measured.
Provider Satisfaction | 6 months
  Clinician experiences and perspectives on satisfaction of the app will be assessed through a study specific satisfaction survey

OTHER OUTCOMES:
Patient Usability | 6 months
  Patient usability will be tracked through the app's data analytics software platform. Study staff will pull data from the data analytics software platform.
Provider usability | 6 months
  Clinician experiences and perspectives on the usability of the Briight app will be assessed a study specific usability survey.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Siminerio, RN, PhD, CDE, Principal Investigator — Professor
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data set used for final analysis will be made available to other researchers who have obtained appropriate regulatory approval
Supporting Information: ICF
Time Frame: Data Set - After publication. ICF - After completing data collection.
Access Criteria: Data set - other researchers will have to request access. ICF will be added to clinicaltrials.gov protocol

REFERENCES:
- [Derived] Krall JS, Childs B, Mehrotra N. Mobile Applications to Support Diabetes Self-Management Education: Patient Experiences and Provider Perspectives. J Diabetes Sci Technol. 2023 Sep;17(5):1206-1211. doi: 10.1177/19322968231174037. Epub 2023 May 10. PMID 37162000